CLINICAL TRIAL: NCT03811886
Title: A Phase I/II Study of Natalizumab as a Single Agent in Children, Adolescents and Young Adults With Recurrent, Refractory or Progressive Pulmonary Metastatic Osteosarcoma
Brief Title: Natalizumab in Recurrent, Refractory or Progressive Pulmonary Metastatic Osteosarcoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No accruals
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1718
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Metastatic Osteosarcoma (pOS)
Keywords: Natalizumab
MeSH Terms: interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Phase I: Natalizumab (Experimental): Traditional 3+3 design escalation of Natalizumab at a weight-based dosing 2mg/kg not to exceed a maximum dose of 300mg
  Phase II treatment to continue if the participant has Complete Response (CR), Partial Response (PR) or Stable Disease (SD) of pOS as defined by RECIST 1.1 criteria after every 3 cycles after the first 6 cycles but not beyond 24 cycles. If the participant has progressive disease after 6 cycles, they will be removed from the study.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Natalizumab is an FDA approved monotherapy for treatment of relapsing forms of MS. It is also indicated for inducing and maintaining clinical response and remission in adult patients with moderately to severely active CD who have had an inadequate response to, or intolerance of, conventional therapies and TNF-α inhibitors.
  Traditional 3+3 escalation of Natalizumab at a weight-based dosing 2mg/kg not to exceed 300mg. If no subjects experience a dose limiting toxicity (DLT), 3 more subjects are enrolled at the next dose of 3mg/kg, not to exceed 300mg. If no subjects experience a DLT, 3 more subjects will be enrolled at the next and final dose of 4mg/kg, not to exceed 300mg.
  Phase II will continue if the subject has Complete Response (CR), Partial Response (PR) or Stable Disease (SD) of pOS, defined by RECIST 1.1 criteria after every 3 cycles after the first 6 cycles but not beyond 24 cycles. If subject has progressive disease after cycle 6, they will be removed from the study.
  Other Names: Tysabri

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Natalizumab in children, adolescent and young adult patients with pulmonary metastatic osteosarcoma (pOS) and to assess clinical response associated with this treatment as well as overall survival.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, proof of concept clinical trial in children, adolescent and young adult patients with unresectable pOS that have progressed, relapsed or are refractory to standard systemic therapy.

All participants will receive the study therapy and there will be dose escalation in a traditional 3 + 3 design during the Phase I study of this trial.

In the Phase II study of the trial, treatment will continue if the subject has Complete Response (CR), Partial Response (PR) or Stable Disease (SD) of pOS after every 3 cycles after the first 6 cycles but not beyond 24 cycles, unless it is judged to be in his/her best interest.

Approximately 3-9 subjects will be enrolled in the phase I part and 10-12 in the phase II part of this trial. Participants will be followed for toxicity for 30 days after treatment has been discontinued or until one of the protocol-defined reasons

This study seeks to evaluate if Natalizumab can be used safely and effectively as immunotherapy in children, adolescent and young adult patients with pOS. Natalizumab is currently Food and Drug Administration (FDA) approved for the treatment of T-cell mediated autoimmune disorders The study team will evaluate the safety and tolerability of Natalizumab as well as the clinical response associated with Natalizumab treatment and evaluate overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female and must be equal to or greater than 5 years of age but less than or equal to 30 years of age at the time of enrollment. No large studies have evaluated the use of Natalizumab in younger pediatric patients, and Natalizumab is currently only FDA approved for adult use; for this reason, children younger than 5 years of age are excluded from this study.
* Subjects must have histologic verification of pOS.
* Subjects must have measurable pulmonary disease or pleural disease per RECIST 1.1 documented by clinical, radiographic and histologic criteria, and have progressed, relapsed or become refractory to conventional therapy.

  -- Subjects despite having peripheral diseases elsewhere outside of pulmonary disease or pleural disease, may be eligible:
  * if these diseases have failed upfront standard therapy AND
  * one or two salvage therapies
* Subjects must have recovered from the acute toxic effects with ≤ Grade 1 as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 of all prior chemotherapy and immunotherapy with the exception of alopecia, anorexia, bone pain, and tumor pain prior to entering this study.
* Myelosuppressive chemotherapy: Must have adequate recovery of counts from previous treatment prior to entry onto this study.
* Monoclonal antibodies: At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody.
* Subjects must have a performance status corresponding to a Karnofsky ≥ 50% for participants > 16 years of age and Lansky ≥ 60 for participants ≤ 16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
* Subjects must have normal organ and marrow function as defined below:
* Adequate bone marrow function defined as:
* Peripheral absolute neutrophil count (ANC) ≥ 750/mcL
* Platelet count ≥ 75,000/mcL (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (may receive packed red blood cell transfusions)
* Adequate liver function defined as:
* Total bilirubin ≤ 1.5 times the upper limit of normal for age
* AST (SGOT) and ALT (SGPT) 2.5 X institutional upper limit of normal
* Serum albumin > 2 g/dL
* Adequate cardiac function defined as:
* Ejection fraction of ≥ 50% by echocardiogram
* Subjects must have the ability to understand and the willingness to sign a written informed consent document if ≥ 18 years of age and an assent document if < 18 years of age. If < 7 years of age, no assent document is required.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment.

* Patients with evidence of osteosarcoma outside of the lungs or pleura.
* Ongoing prior treatment toxicities > Grade 1 according to NCI CTCAE Version 5.0 with the exception of alopecia, anorexia, bone pain and tumor pain.
* Subjects receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Natalizumab.
* Subjects currently on immunosuppressive therapy.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, liver failure, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because Natalizumab crosses the placenta and can increase the risk of spontaneous abortion. There is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with Natalizumab, therefore breastfeeding should be discontinued if the mother is treated with Natalizumab.
* Female participants of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* HIV-positive subjects and HIV-positive subjects on antiretroviral therapy are ineligible because of the risk for developing a lethal infection when treated with immunosuppressive therapy.
* Participants who have or have had progressive multifocal leukoencephalopathy (PML).
* Participants whose pulmonary metastatic disease or pleural disease can be completely surgically resected.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Dosing limiting toxicity | 30 days after end of treatment (1 year)
  Hematologic dose limiting toxicities: Grade 4 neutropenia or thrombocytopenia of > 7 days duration; or myelosuppression that causes a delay of > 8 weeks between treatment courses
  Non-hematologic dose-limiting toxicities: Any Grade 4 non-hematologic toxicity attributable to Natalizumab with the specific exclusion of:
  * Grade 4 nausea and vomiting responding to anti-emetics, alopecia, fatigue and drug related fever
  * Grade 4 fever
  * Any Grade 3 or greater neurologic toxicity
  * Any Grade 3 or greater anaphylaxis
  * Any Grade 2 or greater elevation in transaminases and bilirubin levels
  * Any Grade 4 non-hematologic toxicities (excluding alopecia, nausea and vomiting) that do not resolve to ≤ Grade 1 by 8 weeks following the most recent dose of Natalizumab

SECONDARY OUTCOMES:
Clinical benefit rate | 1 year after start of treatment
  Clinical benefit rate as defined by the number of participants that have Complete Response (CR), Partial Response (PR) or Stable Disease (SD) after 12 cycles
Overall survival measured in months | Up to 3 years
  Overall survival measured in months and summarized using Kaplan-Meier analysis. This will be calculated from the date of registration on-study to the dates of documented evidence of progression or death, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen VanHeyst, DO, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States